CLINICAL TRIAL: NCT04078425
Title: Non Invasive Assessment of Heart Failure
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, salma hamdy mahmoud haridi, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sharidi
Record Dates: First submitted 2019-03-27; First posted 2019-09-06 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: Heart failure; Echocardiography
MeSH Terms: conditions — Heart Failure | interventions — Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HF with preserved EF (Experimental): 50patients of heart failure with preserved ejection fration will receive anti.failure treatment(lanoxin,beta blocker,diuretics) for one month with follow up echocardiography before and after
  Interventions: Drug: Aldosterone Antagonists
- HF with preserved EF recive eplernone (Experimental): 50 patients with heart failure with preserved ejection frationnwill receive traditional anti-failure treatment in addition to aldosterone antagonist (Eplernone) with follow up echocardiography and aldosterone level before and after
  Interventions: Drug: Aldosterone Antagonists

INTERVENTIONS:
Drug: Aldosterone Antagonists — aldosterone antagonist will be applied to patients of heart failure with preserved ejection fraction, level of the drug will be sampled before administration of the drug and follow up will be sampled after one month

SUMMARY:
1. To Identify the role of aldosterone antagonist in patients of heart failure with preserved ejection fraction.
2. Portray the health profile of heart failure patients admitted in internal medicine department either heart failure with reduced ejection fraction or heart failure with preserved ejection fraction.
3. To compare between patients of right and left sided heart failure by biomarkers and parameters of echocardiographgy
4. Vitamin D and its relation to cardiovascular disease and heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is a growing epidemic related to significant morbidity and mortality.

The prevalence of the disease continuously increases due to the ageing population and success in treating cardiovascular diseases that often precede HF.

Lifetime risk of HF is still high with 20-45% and strongly age-dependent . Structural or functional alterations in the heart lead to reduced cardiac output and rising intracardiac pressures.

The resulting HF syndrome comprises typical symptoms such as dyspnoea, ankle swelling and fatigue .

Heart failure is classified into right sided heart failure and left sided heart failure,the later one is classified to HF with reduced EF (HFrEF) involving patients with an EF< 40% and heart failure with preserved ejection fraction (HFpEF) The proportion of HFpEF seems to be slightly lower than that of HFrEF .

For patients presenting with breathlessness, there is a need for a reliable biomarker for the early diagnosis of heart failure. Similarly, there is also a need for better monitoring of patients receiving treatment for heart failure. Non-invasive means such as a biomarker have therefore become useful.

There are many potential biomarkers for heart failure, the investigators will discuss the biomarkers that are available for clinical use in patients with heart failure to further assess prognosis and possibly direct HF therapy.

There is evidence that aldosterone antagonists can oppose the effect of aldosterone in promoting cardiac fibrosis.Furthermore, elevated levels of cardiac aldosterone have been demonstrated in a rat model of hypertensive diastolic HF, and use of the aldosterone antagonist, eplerenone, was associated with attenuation of left ventricular diastolic dysfunction and reduction in left ventricular mass and fibrosis in this model.Thus, aldosterone antagonism has the potential to be a beneficial therapeutic strategy in patients with HFpEF.

Vitamin D has the potential to improve the symptoms ofheart failure (HF) and to modulate the disease,Vitamin D supplementation can reduce blood pressure and improve skeletal muscle function and strength.

Animal studies suggest that active vitamin D down-regulates the renin-angiotensin-aldosterone system (RAAS), reduces retention of salt and water, and reduces myocardial hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosed heart failure dyspnea grade III or IV
2. Heart failure with ejecton fraction ≤40

Exclusion Criteria:

1. Acute coronary syndrome.
2. Active infection
3. Chronic kidney diseased patients
4. Conn's disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Role of aldosterone antagonist in treatment of heart failure | 6months
  To evaluate the effect of aldosterone antagonist on exercise capacity of patients with established and symptomatic HFPEF and to evaluate the effect of aldosterone antagonist on diastolic function (the lateral mitral annular doppler tissue imaging measurments were used for assessment of early diastolic relaxation velocity (E'),ameasure of ventricular relaxation and for calculation of E\E'.